CLINICAL TRIAL: NCT05778487
Title: The Effects of Preoperative Carbohydrate Loading on Elderly Patients Undergoing Orthopaedic Spine Surgery - A CSORN Study
Brief Title: Carbohydrate Loading and Elderly Patients Undergoing Spine Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Horizon Health Network (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HorizonHN
Record Dates: First submitted 2022-06-22; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Diet, Carbohydrate Loading
Keywords: Carbohydrate Loading; Orthopaedics; Elderly; Spine; Cervical; Thoracolumbar; Fusion; Decompression; Discectomy; Gatorade

STUDY DESIGN:
Intervention Model Description: The control group will include retrospectively recruited patients who did not receive preoperative carbohydrate loading, and the carbohydrate (CHO) group will include prospectively recruited patients, who will consume a carbohydrate drink prior to surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Standard of care for dietary instructions only.
  The control group will consist of retrospectively recruited participants who have recently undergone a successful elective spine surgery, and followed the preoperative nutrition standards for their surgery, as outlined by the research institution's fasting dietary guidelines. Recruitment will include the most recent spine surgeries that meet the inclusion criteria and match prospective patient demographics.
- Carbohydrate Group (Experimental): Standard of care for dietary instructions + carbohydrate loading.
  The carbohydrate (CHO) group will consist of prospectively recruited patients scheduled to undergo an elective spine surgery. These participants will also follow the preoperative nutrition standards, however, in addition, they will be instructed to consume 710ml of a simple, commercial carbohydrate sports drink on the day of their procedure up to 2 hours prior to surgery.
  Interventions: Dietary Supplement: Gatorade Thirst Quencher

INTERVENTIONS:
Dietary Supplement: Gatorade Thirst Quencher — Gatorade Thirst Quencher, 710ml (45g of carbohydrates, 6.3% carbohydrates, 25.4kcal/100ml)
  Arms: Carbohydrate Group

SUMMARY:
Carbohydrate loading, the consumption of carbohydrates prior to surgery, is an example of preoperative nutrition that has provided many benefits to surgical patients. Elderly patients (65 years of age and older) represent a large number of spine surgery recipients and due to the unique aspects of aging, proper preoperative nutrition is essential for this patient demographic. The goal of this research study is to determine if preoperative carbohydrate loading provides benefits to elderly patients through decreasing length of stay (LOS) in hospital and reducing perioperative patient adverse events, when undergoing orthopaedic spine surgeries. It is expected that preoperative carbohydrate loading in elderly patients receiving an orthopaedic spine surgery (fusion, decompression, or discectomy) will lead to greater outcomes through decreasing LOS in hospital and reducing perioperative patient adverse events compared to patients who did not receive preoperative carbohydrate loading.

DETAILED DESCRIPTION:
Carbohydrate loading, the consumption of carbohydrates prior to surgery, is an example of preoperative nutrition that has provided many benefits to surgical patients. Because of this, preoperative carbohydrate loading has been included in the Enhanced Recovery After Surgery (ERAS) and Enhanced Recovery Canada (ERC) guidelines across a variety of surgical specialities; however, a gap in the literature remains within the field of orthopaedic surgery, specifically in cervical and thoracolumbar spine surgeries. Elderly patients (65 years of age and older) represent a large number of spine surgery recipients and due to the unique aspects of aging, proper preoperative nutrition is essential for this patient demographic. The goal of this research study is to determine if preoperative carbohydrate loading provides benefits to elderly patients through decreasing length of stay (LOS) in hospital and reducing perioperative patient adverse events, when undergoing orthopaedic spine surgeries. This is an ambispective research study including elderly patients from the Canadian Spine Outcomes and Research Network (CSORN) registry, who have either recently undergone, or are scheduled to undergo, an orthopaedic cervical or thoracolumbar spine surgery (fusion, decompression, or discectomy). The control group will include retrospectively recruited patients, and the carbohydrate (CHO) group will include prospectively recruited patients, who will consume a carbohydrate drink up to 2 hours prior to surgery. Groups will also be matched based on various patient demographic and surgical variables. LOS in hospital and perioperative patient adverse events are the outcome measurements of interest. Patient and surgical variables will also be collected for comparison. It is expected that preoperative carbohydrate loading in elderly patients receiving an orthopaedic spine surgery (fusion, decompression, or discectomy) will lead to greater outcomes through decreasing LOS in hospital and reducing perioperative patient adverse events compared to patients who did not receive preoperative carbohydrate loading.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the age requirement,
* Have either recently undergone, or are scheduled to undergo an elective cervical or thoracolumbar spine surgery, including fusion, decompression, and discectomy procedures.

Exclusion Criteria:

* Potential participants will be excluded if they do not meet the age requirements,
* Have had, or will be having, cervical or thoracolumbar fusion, decompression or discectomy revision surgery,
* Are not able to consume the selected carbohydrate drink,
* Do not consent to participation in the research study,
* Or have diabetes.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Length of Stay (LOS) in Hospital | From the time the patient is admitted to hospital until they are released postoperatively, 0-Maximum hours required.
  How long (hours) are the patients staying in hospital for?

SECONDARY OUTCOMES:
Perioperative Patient Adverse Events | From the time the patient is admitted to hospital until they are released postoperatively, 0-Maximum hours required.
  Do the patients experience any adverse events in hospital such as pain, nausea, vomiting?

CONTACTS AND LOCATIONS:
Overall Officials: Chris Small, MD, Principal Investigator — Canada East Spine Centre
Locations (1):
- Canada East Spine Centre at Saint John Regional Hospital, Saint John, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No
Data cannot be shared publicly because of legal and ethic restrictions. Data from this study are available (contact cescresearch@gmail.com) for researchers who meet the criteria for access to confidential data.

REFERENCES:
- [Background] Kratzing C. Pre-operative nutrition and carbohydrate loading. Proc Nutr Soc. 2011 Aug;70(3):311-5. doi: 10.1017/S0029665111000450. PMID 21781358
- [Background] Yang R, Wolfson M, Lewis MC. Unique Aspects of the Elderly Surgical Population: An Anesthesiologist's Perspective. Geriatr Orthop Surg Rehabil. 2011 Mar;2(2):56-64. doi: 10.1177/2151458510394606. PMID 23569671
- [Background] Altman AD, Helpman L, McGee J, Samouelian V, Auclair MH, Brar H, Nelson GS; Society of Gynecologic Oncology of Canada's Communities of Practice in ERAS and Venous Thromboembolism. Enhanced recovery after surgery: implementing a new standard of surgical care. CMAJ. 2019 Apr 29;191(17):E469-E475. doi: 10.1503/cmaj.180635. No abstract available. PMID 31036609
- [Background] Harsten A, Hjartarson H, Toksvig-Larsen S. Total hip arthroplasty and perioperative oral carbohydrate treatment: a randomised, double-blind, controlled trial. Eur J Anaesthesiol. 2012 Jun;29(6):271-4. doi: 10.1097/EJA.0b013e3283525ba9. PMID 22450530
- [Background] Wainwright TW et al. Consensus statement for perioperative care in total hip replacement and total knee replacement surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Acta Orthop. 2020 Jun;91(3):363. doi: 10.1080/17453674.2020.1724674. Epub 2020 Feb 14. No abstract available. PMID 32056486
- [Background] Debono B, Wainwright TW, Wang MY, Sigmundsson FG, Yang MMH, Smid-Nanninga H, Bonnal A, Le Huec JC, Fawcett WJ, Ljungqvist O, Lonjon G, de Boer HD. Consensus statement for perioperative care in lumbar spinal fusion: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Spine J. 2021 May;21(5):729-752. doi: 10.1016/j.spinee.2021.01.001. Epub 2021 Jan 12. PMID 33444664
- [Background] Baek H, Cho M, Kim S, Hwang H, Song M, Yoo S. Analysis of length of hospital stay using electronic health records: A statistical and data mining approach. PLoS One. 2018 Apr 13;13(4):e0195901. doi: 10.1371/journal.pone.0195901. eCollection 2018. PMID 29652932
- [Background] Singh SM, Liverpool A, Romeiser JL, Miller JD, Thacker J, Gan TJ, Bennett-Guerrero E. A U.S. survey of pre-operative carbohydrate-containing beverage use in colorectal enhanced recovery after surgery (ERAS) programs. Perioper Med (Lond). 2021 May 28;10(1):19. doi: 10.1186/s13741-021-00187-3. PMID 34044894
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Ackerman RS, Tufts CW, DePinto DG, Chen J, Altshuler JR, Serdiuk A, Cohen JB, Patel SY. How Sweet Is This? A Review and Evaluation of Preoperative Carbohydrate Loading in the Enhanced Recovery After Surgery Model. Nutr Clin Pract. 2020 Apr;35(2):246-253. doi: 10.1002/ncp.10427. Epub 2019 Oct 21. PMID 31637778